CLINICAL TRIAL: NCT04136353
Title: DASL-HiCaP: Darolutamide Augments Standard Therapy for Localised Very High-Risk Cancer of the Prostate (ANZUP1801): A Randomised Phase 3 Double-blind, Placebo-controlled Trial of Adding Darolutamide to Androgen Deprivation Therapy and Definitive or Salvage Radiation in Very High Risk, Clinically Localised Prostate Cancer
Brief Title: Darolutamide Augments Standard Therapy for Localised Very High-Risk Cancer of the Prostate
Acronym: DASL-HiCaP
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: University of Sydney (Other)
Collaborators: Australian and New Zealand Urogenital and Prostate Cancer Trials Group (Other); Bayer (Industry); Cancer Trials Ireland (Network); Canadian Cancer Trials Group (Network); Memorial Sloan Kettering Cancer Center (Other); Prostate Cancer Clinical Trials Consortium (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ANZUP1801; U1111-1239-0771 (Other: WHO Universal Trial Number)
Record Dates: First submitted 2019-10-17; First posted 2019-10-23 (Actual); Last update posted 2023-07-28 (Actual); Status verified 2023-07

CONDITIONS: Prostate Cancer
Keywords: clinically localised prostate cancer; very high risk; darolutamide
MeSH Terms: conditions — Prostatic Neoplasms | interventions — darolutamide; Gonadotropin-Releasing Hormone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Darolutamide (Experimental): Darolutamide 600mg (2 x 300mg tablets) twice daily by mouth for 96 weeks, adherence monitored by participant report.
  All participants are treated with an LHRHA for 96 weeks from randomisation and external beam radiation therapy started within 8-24 weeks after randomisation.
  Interventions: Drug: Darolutamide; Drug: Luteinizing Hormone-Releasing Hormone Analog; Radiation: External Beam Radiotherapy
- Placebo (Placebo Comparator): Placebo (2 tablets) twice daily by mouth for 96 weeks, adherence monitored by participant report.
  All participants are treated with an LHRHA for 96 weeks from randomisation and external beam radiation therapy started within 8-24 weeks after randomisation.
  Interventions: Drug: Placebo oral tablet; Drug: Luteinizing Hormone-Releasing Hormone Analog; Radiation: External Beam Radiotherapy

INTERVENTIONS:
Drug: Darolutamide — 2 x 300mg oral tablets twice daily for 96 weeks
  Arms: Darolutamide
Drug: Placebo oral tablet — 2 oral tablets twice daily for 96 weeks
  Arms: Placebo
Drug: Luteinizing Hormone-Releasing Hormone Analog — All participants are to receive standard background therapy with an LHRHA, as per standard of care. The choice of LHRHA is at the discretion of the treating clinician.
Radiation: External Beam Radiotherapy — All participants are to receive standard background therapy with curative-intent RT to the prostate or prostate bed as well as the pelvic lymph nodes using EBRT.

SUMMARY:
The purpose of this study is to determine the effectiveness of darolutamide as part of adjuvant androgen deprivation therapy (ADT) with a luteinising hormone releasing hormone analogue (LHRHA) in men having radiation therapy for localised prostate cancer at very high risk of recurrence.

DETAILED DESCRIPTION:
This trial aims to demonstrate that the use of darolutamide (in addition to standard of care) will be more effective than current standard of care in enhancing the ability of prostate or prostate bed radiation and 96 weeks of androgen suppression in decreasing the number of patients who develop metastases and subsequently die of prostate cancer. Darolutamide is a novel antagonist of the AR with favourable tolerability due to negligible penetration of the blood-brain barrier. Emergence of metastatic disease is the lethal event after local therapy, either with prostatectomy or definitive radiation. Augmenting adjuvant systemic therapy (either ADT or ADT plus docetaxel) with darolutamide has the potential to eradicate micrometastatic disease after either type of local therapy and decrease the death rate from prostate cancer.

This pragmatic design incorporates current standard of care for all patients and the option for docetaxel to be added to ADT. As such, the data will be applicable for all patients with very high risk prostate cancer treated with local therapy and will be the first study incorporating docetaxel use as one of the standard of care options. Even if docetaxel is definitively proven to improve MFS and OS in the adjuvant setting, not all patients will be fit for docetaxel. This will be the first trial that has the potential to build upon current and future advances that may emerge and be the most effective strategy to decrease death rate from prostate cancer in the near term if it further augments docetaxel efficacy in chemo-fit patients.

ELIGIBILITY:
Inclusion Criteria:

1. Men aged 18 years and older, with pathological diagnosis of adenocarcinoma of the prostate
2. EITHER planned for primary RT and judged to be at very high risk for recurrence based on any of the following:

   * Grade Group 5, OR
   * Grade Group 4 AND one or more of the following: clinical T2b-4 OR MRI with seminal vesicle invasion OR extracapsular extension OR PSA* > 20ng/mL, OR
   * Pelvic nodal involvement (involvement of lymph nodes (LNs) at or below the bifurcation of the aorta into the common iliac arteries) defined radiologically as greater than 10mm on short axis using standard CT or MRI, or pathologically confirmed (PSMA PET alone is not considered enough if ≤ 10mm) OR

   Post-radical prostatectomy ≤ 365 days prior to randomisation and planned for RT with PSA* ≥ 0.1 ng/mL that has risen or remained stable (within ≤ 0.05 ng/mL) since a previous level at least 1 week earlier, judged to be at very high risk for recurrence based on any of the following:
   * Grade Group 5, OR
   * Grade Group 4 AND pT3a or higher, OR
   * Pelvic nodal involvement (involvement of LNs at or below the bifurcation of the aorta into the common iliac arteries) defined radiologically as greater than 10mm on short axis using standard CT or MRI, or pathologically confirmed (PSMA PET alone is not considered enough if ≤ 10mm) * This PSA level must be measured within 60 days prior to randomisation. However, if a participant has already commenced endocrine therapy (ET) for prostate cancer, this PSA level must be measured within 180 days prior to commencing ET.
3. Adequate bone marrow function: Haemoglobin ≥ 100g/L, white cell count (WCC) ≥ 4.0x109/L, absolute neutrophil count (ANC) ≥ 1.5x109/L and platelets > 100 x 109/L
4. Adequate liver function: alanine aminotransferase (ALT) < 2 x upper limit of normal (ULN) and total bilirubin < 1.5 x ULN, (or if total bilirubin is between 1.5 - 2 x ULN, they must have a normal conjugated bilirubin)
5. Adequate renal function: calculated creatinine clearance > 30 mL/min (Cockroft-Gault)
6. Eastern Cooperative Oncology Group (ECOG) performance status of 0 - 1
7. Study treatment both planned and able to start within 7 days after randomisation
8. Willing to complete health-related quality of life (HRQL) questionnaires UNLESS is unable to complete because of literacy or limited vision
9. Willing and able to comply with all study requirements, including standard of care treatment such as EBRT, timing and/or nature of required assessments
10. Signed, written informed consent

    Exclusion Criteria:
11. Prostate cancer with predominant non-adenocarcinoma features (sarcomatoid or spindle cell or neuroendocrine small cell or squamous cell components or other non-adenocarcinoma)
12. Involvement of LNs by conventional CT imaging superior to the common iliac artery bifurcation, and/or outside the pelvis (distant LNs). LN involvement is defined by histopathological confirmation, or by a short axis measurement > 10mm on standard imaging (CT or MRI, but not PET).
13. Evidence of metastatic disease. Minimum imaging requirements to exclude metastatic disease are diagnostic quality imaging of both the pelvis and the abdomen (CT or MRI), chest (CXR or CT), and a whole body radioisotope bone scan (WBBS).

    * If endocrine therapy (ET) had not started, imaging must be within 60 days prior to randomisation.
    * If ET has been started, imaging must have been performed no more than 60 days prior to starting ET and no more than 30 days after starting ET and prior to randomisation.
14. PSA > 100 ng/mL at any time
15. Any prior use of new generation potent AR inhibition (abiraterone, enzalutamide, apalutamide, darolutamide or similar agents).
16. Prior endocrine therapy for prostate cancer except for the following which are allowed:

    * (i) LHRHA and/or (ii) a first-generation nonsteroidal antiandrogen (NSAA) are allowed if commenced no more than 90 days before randomisation. If an NSAA has been used, it must be stopped before starting study treatment with darolutamide/placebo; and
    * Prior use of 5-alpha reductase inhibitor is allowed and if used it must be stopped before starting study treatment with darolutamide/placebo
17. Bilateral orchidectomy
18. Prior pelvic brachytherapy or other radiotherapy that would result in an overlap of radiotherapy fields that would preclude the required RT
19. History of

    * Loss of consciousness or transient ischemic attack or stroke within 6 months prior to randomisation, or
    * Significant cardiovascular disease within 6 months prior to randomisation: including myocardial infarction, unstable angina, congestive heart failure (NYHA grade II or greater), ongoing arrhythmias of Grade > 2 (CTCAE v5.0), thromboembolic events (e.g. deep vein thrombosis, pulmonary embolism), coronary artery bypass graft. Chronic stable atrial fibrillation on stable anticoagulant therapy is allowed.
20. Known gastrointestinal (GI) disease or GI procedure that could interfere with the oral absorption or tolerance of darolutamide, including difficulty swallowing tablets
21. History of another malignancy within 5 years prior to randomisation except for those malignancies treated with curative intent with a predicted risk of relapse of less than 10% including but not limited to non-melanoma carcinoma of the skin; or adequately treated, non-muscle-invasive urothelial carcinoma of the bladder (i.e. Tis, Ta and low grade T1 tumours). All such cases with a history of malignancy within the last 5 years are to be discussed with study team before randomisation. Melanoma in-situ and other adequately treated in-situ neoplasms are not considered malignancies for the purposes of eligibility assessment.
22. Concurrent illness, including severe infection that might jeopardise the ability of the participant to undergo the procedures outlined in this protocol with reasonable safety (HIV infection is not an exclusion criterion if it is controlled with anti-retroviral drugs that are unaffected by concomitant darolutamide)
23. Presence of any psychological, familial, sociological or geographical condition potentially hampering compliance with the study protocol and follow-up schedule, including alcohol dependence or drug abuse
24. Patients who are sexually active with women of child-bearing potential and not willing/able to use medically acceptable and highly effective forms of contraception during study treatment and for at least 4 weeks after completion of study treatment. Contraception must include:

    * Condom use (also required if sexual partner is pregnant), and
    * Additional birth control with low failure rate (less than 1% per year) when used consistently and correctly. E.g. combined (oestrogen and progestogen containing) hormonal contraception associated with inhibition of ovulation (oral, intravaginal, transdermal), progestogen-only hormonal contraception associated with inhibition of ovulation (oral, injectable, implantable), intrauterine device (IUD), intrauterine hormone-releasing system (IUS), bilateral tubal occlusion, vasectomised partner, true sexual abstinence.

    True sexual abstinence will only be an acceptable form of contraception when this is in line with the preferred and usual lifestyle of the subject. Periodic abstinence (e.g., calendar, ovulation, symptothermal, post-ovulation methods), declaration of abstinence for the duration of exposure to study treatment, and withdrawal are not acceptable methods of contraception.
25. Participation in other clinical trials of investigational agents for the treatment of prostate cancer or other diseases
26. Major surgery within 21 days prior to randomisation
27. Patients with history of hypersensitivity to the study treatment

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1100 (Actual)
Dates: Start 2020-03-31 (Actual); Primary Completion 2028-01-31 (Estimated); Study Completion 2028-07-31 (Estimated)

PRIMARY OUTCOMES:
Metastasis-free survival | Through study completion, an average of 5 years
  Evidence of metastases includes findings on WBBS or CT or MRI (as reported by the site investigator) that are either characteristic of metastatic prostate cancer, and/or confirmed by other test results e.g. cytology or histopathology.

SECONDARY OUTCOMES:
Overall survival | Through study completion, an average of 5 years
  Overall survival is defined as the interval from the date of randomisation to date of death from any cause, or the date of last known follow-up alive.
Prostate cancer-specific survival | Through study completion, an average of 5 years
  Prostate cancer-specific survival is defined as the interval from the date of randomisation to the date of last known follow-up alive, or the date of death from prostate cancer. Deaths from other causes will be summarised.
PSA-progression free survival | Through study completion, an average of 5 years
  For participants who receive definitive radiotherapy (i.e. without radical prostatectomy), PSA progression is defined by the Phoenix criteria (requires confirmation by a repeat PSA performed at least 3 weeks later). For participants who have undergone a radical prostatectomy, an increase in PSA of >0.2 ng/mL above the nadir would be considered PSA progression (requires confirmation by a repeat PSA performed at least 3 weeks later).
Time to subsequent hormonal therapy | Through study completion, an average of 5 years
  Time to subsequent hormone therapy is the interval from randomisation to the first date that endocrine therapy is recommenced or changed for the treatment of recurrent (or progressive) prostate cancer.
Time to castration-resistance | Through study completion, an average of 5 years
  Defined according to the PCWG3 criteria. If a participant has radiographic progression without serological progression, this will also be deemed castration resistant prostate cancer
Frequency and severity of adverse events (CTCAE v5.0, RTOG/EORTC acute/late radiation morbidity criteria) | Approximately 12-weekly for 2 years from randomisation until 30 days after the last dose of study treatment.
  Safety reporting will describe the frequency and severity of AEs. The CTCAE v5.0 will be used to classify and grade the intensity of AEs occurring until 30 days after the last dose of study treatment. The RTOG/EORTC Scoring Criteria will be used to assess morbidities related to radiation therapy (RT) until 6 years after randomisation. Acute AEs are those occurring within 90 days after starting RT, and will be classified and graded according to the RTOG/EORTC Acute Radiation Morbidity Scoring Criteria. Late AEs are those occurring more than 90 days after starting RT, and will be classified and rated according to the RTOG/EORTC Late Radiation Morbidity Scoring Schema.
Health-related quality of life | Through study completion, an average of 5 years
  EORTC Core Quality of Life Questionnaire (QLQC-30). Importance of quality of life issues are assessed using a four-point scale (1 = not at all, 4 = very much)
  EORTC Quality of Life Questionnaire for Prostate Cancer (PR-25). Importance of quality of life issues are assessed using a four-point scale (1 = not at all, 4 = very much)
  Euroqol 5 item preference-based measure of health (EQ-5D-5L), comprising 5 questions with a score from 1 to 5 each and a visual analogue scale from 0 to 100.
Fear of cancer recurrence | Through study completion, an average of 5 years
  Using the Fear of Cancer Recurrence Inventory (FCRI), a 42-item questionnaire with scores of 0 (never/not at all) - 4 (all the time/a great deal) for each.

CONTACTS AND LOCATIONS:
Overall Officials: Christopher Sweeney, Study Chair — Dana-Farber Cancer Institute and Harvard Medical School; Tamim Niazi, Study Chair — Jewish General Hospital and McGill University
Locations (93):
- United States (19):
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - Dana Farber Cancer Institute - St. Elizabeth's, Brighton, Massachusetts
  - Lahey Hospital and Medical Center, Burlington, Massachusetts
  - Dana Farber Cancer Institute - Milford, Milford, Massachusetts
  - XCancer Omaha/Urology Cancer Center, Omaha, Nebraska
  - Memorial Sloan Kettering Basking Ridge, Basking Ridge, New Jersey
  - New Jersey Urology Saddle Brook, Clifton, New Jersey
  - Memorial Sloan Kettering Monmouth, Middletown, New Jersey
  - Memorial Sloan Kettering Bergen, Montvale, New Jersey
  - New Jersey Urology Voorhees, Voorhees Township, New Jersey
  - New Mexico Oncology and Hematology Specialists, Albuquerque, New Mexico
  - Memorial Sloan Kettering Commack, Commack, New York
  - Memorial Sloan Kettering Westchester, Harrison, New York
  - New York University Langone Long Island, Mineola, New York
  - New York University Langone Medical Center, New York, New York
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - Memorial Sloan Kettering Nassau, Uniondale, New York
  - Dayton Physicians Network, Kettering, Ohio
  - Seattle Cancer Care Alliance, Seattle, Washington
- Australia (32):
  - Border Medical Oncology Research Unit, Albury, New South Wales
  - Gosford Hospital, Gosford, New South Wales
  - GenesisCare Newcastle, Newcastle, New South Wales
  - Calvary Mater Newcastle, Newcastle, New South Wales
  - Shoalhaven District Memorial Hospital, Nowra, New South Wales
  - St Vincent's Public Hospital, Sydney, New South Wales
  - Prince of Wales Hospital, Sydney, New South Wales
  - Chris O'Brien Lifehouse, Sydney, New South Wales
  - Northern Cancer Institute, Sydney, New South Wales
  - Sydney Adventist Hospital, Sydney, New South Wales
  - Liverpool Hospital, Sydney, New South Wales
  - St George Hospital, Sydney, New South Wales
  - Campbelltown hospital, Sydney, New South Wales
  - Wollongong Hospital, Wollongong, New South Wales
  - ROPART, Brisbane, Queensland
  - Royal Brisbane and Women's Hospital, Herston, Queensland
  - Icon Cancer Centre, Southport, Queensland
  - Townsville Hospital, Townsville, Queensland
  - Princess Alexandra Hospital, Woolloongabba, Queensland
  - Ashford Cancer Centre Research, Kurralta Park, South Australia
  - Icon Cancer Centre Hobart, Hobart, Tasmania
  - Royal Hobart Hospital, Hobart, Tasmania
  - Peter MacCallum Cancer Centre - Bendigo Campus, Bendigo, Victoria
  - Peter MacCallum Cancer Centre (Moorabbin Campus), Bentleigh East, Victoria
  - Box Hill Hospital, Box Hill, Victoria
  - GenesisCare Cabrini (Gandel Wing), Cabrini Hospital Malvern, Malvern, Victoria
  - Peter MacCallum Cancer Centre, Melbourne, Victoria
  - The Alfred Hospital, Melbourne, Victoria
  - Sunshine Hospital, St Albans, Victoria
  - Latrobe Regional Hospital, Traralgon, Victoria
  - Fiona Stanley Hospital, Murdoch, Western Australia
  - Sir Charles Gairdner Hospital, Nedlands, Western Australia
- Canada (20):
  - Cross Cancer Institute, Edmonton, Alberta
  - BC Cancer Agency (BCCA) Fraser Valley, Surrey, British Columbia
  - Western Manitoba Cancer Centre - Prairie Mountain Health, Brandon, Manitoba
  - CancerCare Manitoba, Winnipeg, Manitoba
  - Regional Health Authority B, Zone 2 Saint John Regional Hospital, Saint John, New Brunswick
  - Dr. H. Bliss Murphy Cancer Centre, St. John's, St. John's, Newfoundland and Labrador
  - Kingston Health Sciences Centre, Kingston, Ontario
  - Queen Elizabeth II Health Sciences Centre, London, Ontario
  - Sault Area Hospital - Algoma District Cancer Program, Sault Ste. Marie, Ontario
  - Ottawa Hospital Research Institute, Toronto, Ontario
  - Odette Cancer Centre - Sunnybrook Hospital, Toronto, Ontario
  - Princess Margaret Cancer Centre, Toronto, Ontario
  - Centre Integre de Sante et de Services Sociaux de la Monteregie Centre, Greenfield Park, Quebec
  - Jewish General Hospital, Montreal, Quebec
  - Centre Hospitalier de l'Universite de Montreal, Montreal, Quebec
  - Hôtel-Dieu de Québec, Québec, Quebec
  - Centre Hospitalier Universitaire de Sherbrooke, Sherbrooke, Quebec
  - Allan Blair Cancer Centre, Regina, Saskatchewan
  - Saskatoon Cancer Centre, Saskatoon, Saskatchewan
  - Centre Hospitalier Regional de Trois-Rivieres, Québec
- Ireland (9):
  - St. Luke's Hospital, Rathgar, Dublin 6
  - Cork University Hospital, Cork
  - Bon Secours Hospital Cork in association with UPMC Hillman Centre, Cork
  - Mater Misericordiae University Hospital, Dublin
  - Mater Private Dublin, Dublin
  - St Luke's Radiation Oncology Network at St James's Hospital, Dublin
  - Beacon Private Hospital Dublin, Dublin
  - Tallaght University Hospital, Dublin
  - Galway University Hospital, Galway
- New Zealand (3):
  - Auckland City Hospital, Auckland
  - Christchurch Hospital, Christchurch
  - Palmerston North Hospital, Palmerston North
- United Kingdom (10):
  - Aberdeen Royal Infirmary, Aberdeen
  - William Harvey Hospital, Ashford
  - Royal United Hospital Bath, Bath
  - Belfast City Hospital, Belfast
  - Kent and Canterbury Hospital, Canterbury
  - Western General Hospital, Edinburgh
  - Beatson West of Scotland Cancer Centre, Glasgow
  - Guy's and St Thomas Hospital, London
  - Royal Marsden Hospital, London
  - Nottingham University Hospitals NHS Trust - Nottingham City Hospital, Nottingham